CLINICAL TRIAL: NCT02312882
Title: Tofacitinib for the Treatment of Alopecia Areata and Its Variants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anthony Oro, Principle Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31790ORO; IRB-31790 (Other: Stanford University)
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Alopecia Areata; Alopecia Totalis; Alopecia Universalis
MeSH Terms: conditions — Alopecia Areata; Alopecia universalis | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tofacitinib (Experimental): Participants will receive tofacitinib for 3 months.
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — Tofacitinib 5 mg tablet taken by mouth twice a day.
  Other Names: Xeljanz; Jakvinus

SUMMARY:
The purpose of this study is to investigate the ability of tofacitinib citrate, a Janus kinase inhibitor, to generate hair regrowth in patients with moderate to severe alopecia areata and its variants.

DETAILED DESCRIPTION:
This study is an open-label pilot study. Participants will be treated with oral tofacitinib for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Diagnosis of alopecia areata with >50% scalp involvement, alopecia totalis, or alopecia universalis
* Hair loss present for at least 6 months
* No treatment for alopecia areata in past 2 months
* No evidence of hair regrowth
* Females of childbearing potential must use birth control while taking the medication and there must be a negative pregnancy test documented prior to starting the medication
* Fluent in spoken and written English

Exclusion Criteria:

* Age <18 years old
* Patients have received treatment known to affect alopecia areata within 2 months of enrolling in the study
* Patients with a history of malignancy (except history of successfully treated basal cell or squamous cell carcinoma of the skin)
* Patients known to be HIV or hepatitis B or C positive
* Patients with positive tuberculin skin test or positive QuantiFERON TB test
* Patients with leukopenia or anemia
* Patients with renal or hepatic impairment
* Patients with peptic ulcer disease
* Patients taking immunosuppressive medications, including but not limited to prednisone, methotrexate, mycophenolate mofetil, azathioprine, tacrolimus, cyclosporine, or TNH-alpha inhibitors
* Women of childbearing potential who are unable or unwilling to use birth control while taking the medication
* Women who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony E Oro, M.D., Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- [Result] Kennedy Crispin M, Ko JM, Craiglow BG, Li S, Shankar G, Urban JR, Chen JC, Cerise JE, Jabbari A, Winge MC, Marinkovich MP, Christiano AM, Oro AE, King BA. Safety and efficacy of the JAK inhibitor tofacitinib citrate in patients with alopecia areata. JCI Insight. 2016 Sep 22;1(15):e89776. doi: 10.1172/jci.insight.89776. PMID 27699252

RESULTS

PARTICIPANT FLOW:
Groups:
- Tofacitinib: Tofacitinib (5 mg tablet taken by mouth twice a day) for 3 months.
Period: Overall Study
Arm/Group | Tofacitinib
Started | 40
Completed | 36
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: Participants who completed the protocol are included in the analysis.
Groups:
- Treatment Arm: Tofacitinib (5 mg tablet taken by mouth twice a day) for 3 months.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: years] | 37 [19 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Severity of Alopecia Tool (SALT) Score
Description: SALT score range is from 0 (no hair loss) to 100 (100% hair loss). Positive percent change from baseline corresponds to reduction in SALT score.
Time Frame: 0 and 3 months
Measure: Median (Full Range); unit: Percent change
Arm/Group | Treatment Arm
Number analyzed (Participants) | 36
Percent change | 30.7 [0 to 87.4]
Statistical Analysis 1: Comparison: Treatment Arm; Test type: Other; p < 0.0001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Treatment Arm
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 18/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=40)
Abdominal pain (Gastrointestinal disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 2
Conjunctivitis (Eye disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Dry eyes (Eye disorders) | 1
Fatigue (General disorders) | 2
Folliculitis (Skin and subcutaneous tissue disorders) | 1
Headache (Nervous system disorders) | 2
Hot flashes (Endocrine disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Numbness (General disorders) | 1
Paronychia (Infections and infestations) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 4
Urinary tract infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes